CLINICAL TRIAL: NCT03029299
Title: Implementation Assessment and Clinical Utility of the FilmArray® Respiratory Panel (RP) EZ in a CLIA-waived Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioFire Diagnostics, LLC (Industry)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: DX-SDY-031041
Record Dates: First submitted 2017-01-14; First posted 2017-01-24 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Respiratory Tract Infections
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (No Intervention): Subjects receive standard of care testing as determined by the clinician.
- Intervention (Experimental): Subjects are tested using the FilmArray RP EZ and the results are provided to the clinician for use in determination of patient care (along with any other clinician-ordered testing)
  Interventions: Device: FilmArray RP EZ

INTERVENTIONS:
Device: FilmArray RP EZ — Patients in the intervention arm will be tested with the FilmArray RP EZ and the results of the test will be provided to the treating clinician
  Arms: Intervention

SUMMARY:
BioFire Diagnostics, LLC (BioFire; a bioMerieux company), has developed a multiplexed molecular-based in vitro diagnostic platform for infectious disease testing known as the FilmArray. The FilmArray Respiratory Panel (RP) EZ is a test designed for use with the FilmArray 2.0 EZ Configuration instrument that identifies common bacterial and viral microorganisms associated with respiratory tract infections from a nasopharyngeal swab (NPS) specimen collected in viral transport media (VTM). The RP EZ was granted CLIA-waived classification by the FDA in October 2016 and is the first highly-multiplexed molecular test to receive this designation.

The purpose of this study is to measure patient outcomes following implementation of the RP EZ test and to also gather data about physician office workflow and user interactions with the device. These data will be used to understand how the adoption of such tests may influence patient care in the CLIA-waived setting.

DETAILED DESCRIPTION:
The FilmArray RP EZ may offer improvements over conventional CLIA-waived testing for respiratory infections. Molecular-based testing provides increased sensitivity and specificity relative to current clinical reference methods and multiplexed panels offer a greater breadth of organism identification and diagnostic yield than is available using standard methods available in the CLIA-waived setting. Because of these attributes, the results from this test have the potential to enable clinicians to more accurately diagnose and treat respiratory illness.

It is hypothesized that the sensitive, specific, and comprehensive results provided by FilmArray RP EZ will allow clinicians to more rapidly diagnose respiratory illness and implement appropriate therapy, as well as provide subjects with appropriate expectations about their course of illness.

This interventional clinical trial that will be initiated during the 2016-2017 respiratory illness season to measure the utility of FilmArray RP EZ when implemented in an outpatient care setting. At least three different outpatient or urgent care clinics within the UCLA Health system will be selected for participation. Subjects will be randomized into two groups within each site. The control group will receive standard of care according to the subject's provider's determination. The intervention group will receive testing with FilmArray RP EZ.

Outcome measures will include (but are not limited to) total healthcare costs, antimicrobial prescription rates, timeliness, and appropriateness of therapy, clinician attitudes towards laboratory test capabilities, and subject satisfaction with their healthcare encounter.

As specimens will be collected specifically for this research study, written informed consent, assent, and/or parental permission will be obtained from all study participants.

ELIGIBILITY:
Inclusion Criteria:

* Subject presents with signs/symptoms of respiratory infection including but not limited to fever, cough, sore throat, runny nose, myalgia, headache, chills, or fatigue.
* Subject provides written informed consent/assent/parental permission
* Willing and able to provide NPS specimen

Exclusion Criteria:

* Subject is unable to provide consent/assent/parental permission
* Children whose legal guardian is not available to give permission
* Unable/unwilling to provide NPS specimen
* Non-English speaking

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Time duration from initial visit to receipt of appropriate therapy | through study completion, an average of one year
  Time to appropriate therapy as measured in days compared between intervention and control arms.

SECONDARY OUTCOMES:
Satisfaction scores | through study completion, an average of one year
  Subject and clinician satisfaction with healthcare encounter as measured on 4 point preference scale (highly satisfied, satisfied, dissatisfied, highly dissatisfied) and compared between intervention and control arms
Total healthcare costs | through study completion, an average of one year
  Comparison of total healthcare costs measured in dollars for patients in Control vs Intervention arm

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No